CLINICAL TRIAL: NCT05663606
Title: Glycemic Outcomes and Diabetes Distress in Children With Type 1 Diabetes Aged 9-13 Years Using Happy Bob -Application
Brief Title: Happy Bob App in 9-13 Year-old Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: DexCom, Inc. (Industry)
Responsible Party: Principal Investigator, Tero Varimo, MD, PhD, Principal Investigator, Pediatric Endocrinologist, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OUS-2022-028
Record Dates: First submitted 2022-12-02; First posted 2022-12-23 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Type1diabetes
Keywords: Type 1 diabetes; Continuous glucose monitoring; Gamification; Time in Range
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: prospective, randomized, controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Happy Bob Arm (Active Comparator): Subjects, who are using Happy Bob App in addition to CGM
  Interventions: Combination Product: Happy Bob; Device: CGM
- Controls (Placebo Comparator): Subjects, who are using CGM only
  Interventions: Device: CGM

INTERVENTIONS:
Combination Product: Happy Bob — Application, which gives stars when subject reachs Time In Range
  Arms: Happy Bob Arm
Device: CGM — Dexcom CGM

SUMMARY:
The purpose of the study is to evaluate the effectiveness of the Happy Bob -application on glycemic control in children aged 9-13 years with type 1 diabetes. Additionally, investigators evaluate the perceived burden on the diabetes treatment to families during the Happy Bob use, compared to conventional treatment (diabetes distress).

This is a prospective, randomized, controlled study where primary endpoint is the change in time-in-range (TIR, 3.9-10 mmol/l) after Happy Bob application initiation. Secondary endpoints are HbA1c, time below range (TBR, <3.9 mmol/l), time above range (TAR, >10 mmol/l), mean sensor glucose (SG), standard deviation of SG, coefficient of variation (CV, SD/SGx100 (%)), number of boluses and diabetes distress evaluated by PAID (Problem Areas In Diabetes for parents and children/youth). A sample size of 40 subjects (20 in each groups, and assumed drop-out rate of 10%) would provide the trial with 80% power and type 1 error rate of 0.05 with the following assumption: 7% higher TIR during Happy Bob -use compared to conventional treatment with continuous glucose monitoring (CGM), with a standard deviation of 7.5% (based on Happy Bob marketing study).

The inclusion criteria are 1) Type 1 diabetes diagnosis more than 6 months ago 2) Age 9-13 years and prepubertal 3) capability to use Happy Bob -app and continuous glucose monitoring (CGM). The exclusion criteria are psychiatric diagnosis and other conditions, which in the opinion of the investigator would put the participant at risk during the trial.

The study includes 6 months study time with 2 standard outpatient clinic visits.

DETAILED DESCRIPTION:
The study will be conducted at pediatric diabetes outpatient clinics of Helsinki University Hospital (New Children's Hospital, Jorvi Hospital, Lohja Hospital, Porvoo Hospital and Raasepori Hospital).

The study protocol is explained to the participants (9-13 -year-old children) and their guardian(s). Informed consent from participants' caregivers and participants will be taken by investigators, clinicians or diabetes nurses. The investigator or his/her representative will explain the nature of the study to the patient and parents, and answer all questions regarding the study. Prior to any study-related screening procedures, the informed consent statement will be reviewed and signed and dated by the participant's caregiver.

The participants are using their usual diabetes treatment (multiple daily injections, MDI, or continuous subcutaneous insulin infusion, CSII) with Dexcom™ G6 (Dexcom Inc., San Diego, CA) CGM during the study period and will get instructions for insulin treatment from their diabetes nurses/doctors as usual. Study group will also use Happy Bob application, which takes data from Dexcom CGM system, and gives a user a star, whenever he/she is within target area, measured every five minutes. The more stars patients get, the better the score is. Happy Bob is not a medical device, and it does not give any instructions on how to dose insulin. The use of CGM is familiar to subjects and their families, since every patient is already using some CGM before the study. If Dexcom CGM is not the CGM device patients uses normally, the instructions for the use is given by study nurses either remotely (video appointment) or during outpatient clinic group visit.

The instruction for the Happy Bob use is given by study nurse in groups, either remotely (video appointment) or in outpatient clinic group visit.

The used CGM is Dexcom G6 sensor, which is integrated to Happy Bob -app. It measures the glucose level in the subcutaneous tissue. The CGM sensor connects to a transmitter that sends the glucose data to patients phone (Dexcom app) and receiver device. The sensor is worn for 10 days and then replaced with a new one by the patients' caregivers. The CGM data are collected from Glooko® Therapy management software, which is in clinical use at Helsinki University Hospital. The data from CGM is downloaded either by caregivers or diabetes nurse at diabetes clinic.

Glycated haemoglobin (HbA1c, mmol/mol) (Afinion2™, Abbott) is measured by a diabetes nurse from fingertip as point of care test. The Diabetes Distress is evaluated by a standardized questionnaire (PAID) in run-in phase and at 6 months visit.

The study includes a starting visit, during which Happy Bob and Dexcom G6 CGM is started and patient's normal outpatient clinic visits in 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes diagnosis more than 6 months ago
* Age 9-13 years
* Prepubertal
* Capability to use Happy Bob -app and continuous glucose monitoring (CGM)

Exclusion Criteria:

* Psychiatric diagnosis and other conditions, which in the opinion of the investigator would put the participant at risk during the trial.

Ages: 9 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
TIR | 6 months
  Change in time in range, 3.9-10 mmol/l (%)

SECONDARY OUTCOMES:
TBR | 6 months
  change in time below range (<3.9 mmol), %
TAR | 6 months
  change in time above range (>10.0 mmol), %
SG | 6 months
  change in mean sensor glucose value (SG) (mmol/l)
SD | 6 months
  change in standard deviation of sensor glucose values (mmol/l)
CV | 6 months
  change in coefficient of variation of sensor glucose values (SG/SDx100),%
Boluses | 6 months
  number of boluses/day (lowest 0, highest not defined)
Diabetes distress | 6 months
  PAID (problem areas in diabetes) score: 0-100, higher score indicates more burden
HbA1c | 6 months
  glycated haemoglobin, mmol/mol

IPD SHARING:
Plan to Share IPD: No